CLINICAL TRIAL: NCT02639494
Title: Self-Centering Guide Catheter Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: S2360
Record Dates: First submitted 2015-12-17; First posted 2015-12-24 (Estimated); Results first posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Self-Centering Guide Catheter (Experimental): Subjects who provided written informed consent and an attempt is made to insert the Self-Centering Guide Catheter into the subject's femoral artery.
  Interventions: Device: Self-Centering Guide Catheter

INTERVENTIONS:
Device: Self-Centering Guide Catheter

SUMMARY:
An evaluation of the feasibility of using the Self-Centering Guide Catheter to deliver a guide wire across a stenotic native aortic valve into the left ventricle.

DETAILED DESCRIPTION:
A prospective, open-label, single-arm feasibility study evaluating the Self-Centering Guide Catheter. All subjects who are candidates for transcatheter aortic valve replacement (TAVR) of a native valve with a transcatheter aortic valve that is introduced percutaneously via the femoral artery using conventional catheterization techniques will be evaluated for enrollment in this study. The Self-Centering Guide Catheter is intended to facilitate delivery of a guidewire across a stenotic native aortic valve and into the left ventricle.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age.
* Subject (or legal guardian) understands the study requirements and the treatment procedures and provides written informed consent before any study-specific tests or procedures are performed.
* Subject is eligible for and is an acceptable candidate for transcatheter aortic valve replacement of a stenotic (aortic valve area ≤1 cm2, aortic jet velocity ≥4.0 m/s, or mean gradient ≥40 mmHg) native valve with a transcatheter aortic valve that is introduced percutaneously via the femoral artery using conventional catheterization techniques.

Exclusion Criteria:

* Subject has known hypersensitivity to the components of the device (e.g., polyether block amide, fluoropolymers, nickel, platinum, tantalum, titanium).
* Subject has a pre-existing prosthetic aortic valve.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05-12 (Actual); Primary Completion 2016-10-06 (Actual); Study Completion 2016-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Gulati, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Self-Centering Guide Catheter: Subjects who provided written informed consent and an attempt was made to insert the Self-Centering Guide Catheter into the subject's femoral artery.
Period: Overall Study
Arm/Group | Self-Centering Guide Catheter
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Self-Centering Guide Catheter
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.0 (9.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Self-Centering Guide Catheters Successfully Used to Deliver a Guide Wire Through the Self-Centering Guide Catheter Across the Stenotic Native Aortic Valve Into the Left Ventricle
Description: This outcome will be assessed via physician determination and will be recorded in the case report form.
Time Frame: Through study completion, up to 72 hours post-procedure
Population: 20 patients were treated with 23 devies
Measure: Count of Units; unit: Device
Units Other Than Participants: Device
Arm/Group | Self-Centering Guide Catheter
Number analyzed (Participants) | 20
Number analyzed (Device) | 23
Device | 18

2. Other Pre Specified Outcome: Time From Insertion of the Self-Centering Guide Catheter Into the Body to Successful Placement of a PTFE-coated Guidewire Across the Stenotic Native Aortic Valve
Time Frame: Through study completion, up to 72 hours post-procedure
Population: A guide wire was delivered through the self-centering guide catheter in 18/20 patients.
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Self-Centering Guide Catheter
Number analyzed (Participants) | 18
minutes | 3.8 [2.7 to 4.8]

3. Other Pre Specified Outcome: Time From Insertion of the Self-Centering Guide Catheter Into the Body to Removal of the Self-Centering Guide Catheter From the Body
Time Frame: Through study completion, up to 72 hours post-procedure
Population: A guide wire was delivered through the self-centering guide catheter in 18/20 patients. In total 23 devices were used.
Measure: Mean (95% Confidence Interval); unit: minutes
Units Other Than Participants: Devices
Arm/Group | Self-Centering Guide Catheter
Number analyzed (Participants) | 18
Number analyzed (Devices) | 23
minutes | 6.6 [4.4 to 8.8]

4. Other Pre Specified Outcome: Number of Attempts Made to Cross the Stenotic Native Aortic Valve With a PTFE-coated Guidewire
Time Frame: Through study completion, up to 72 hours post-procedure
Measure: Mean (95% Confidence Interval); unit: Attempts
Units Other Than Participants: Device
Arm/Group | Self-Centering Guide Catheter
Number analyzed (Participants) | 20
Number analyzed (Device) | 23
Attempts | 5.1 [3.2 to 7.0]

5. Other Pre Specified Outcome: Successful Recapture of the Distal Self-centering Basket of the Device Into the Guide and Withdrawal of the Self-Centering Guide Catheter Through the Guide System
Description: The outcome measure of successful recapture of the distal self-centering basket of the device into the guide and withdrawal of the Self-Centering Guide Catheter through the guide system will be assessed via physician assessment of the self-centering basket recapture and will be recorded in the case report form.
Time Frame: Through study completion, up to 72 hours post-procedure
Measure: Count of Units; unit: Device
Units Other Than Participants: Device
Arm/Group | Self-Centering Guide Catheter
Number analyzed (Participants) | 20
Number analyzed (Device) | 23
Device | 23

6. Other Pre Specified Outcome: Number of Self-Centering Guide Catheters With Device Success
Description: Device success is defined as successful delivery of a guide wire through the Self-Centering Guide Catheter across the stenotic native aortic valve into the left ventricle and successful recapture of the distal self-centering basket of the device into the guide and withdrawal of the Self-Centering Guide Catheter through the guide system. This outcome will be assessed via physician determination and will be recorded in the case report form.
Time Frame: Through study completion, up to 72 hours post-procedure
Measure: Count of Units; unit: Device
Units Other Than Participants: Device
Arm/Group | Self-Centering Guide Catheter
Number analyzed (Participants) | 20
Number analyzed (Device) | 23
Device | 18

7. Other Pre Specified Outcome: Number of Participants With Stroke
Time Frame: 72 hours post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Centering Guide Catheter
Number analyzed (Participants) | 20
Participants | 0

8. Other Pre Specified Outcome: Number of Participants With Cardiac Tamponade
Time Frame: 72 hours post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Centering Guide Catheter
Number analyzed (Participants) | 20
Participants | 0

9. Other Pre Specified Outcome: Death, All-cause, Cardiovascular, and Non-cardiovascular
Time Frame: 72 hours post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Centering Guide Catheter
Number analyzed (Participants) | 20
Participants | 0

10. Other Pre Specified Outcome: Any Device-related Adverse Event
Time Frame: 72 hours post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Centering Guide Catheter
Number analyzed (Participants) | 20
Participants | 0

11. Other Pre Specified Outcome: Any Adverse Event Occurring While the Self-Centering Guide Catheter is in the Subject
Time Frame: 72 hours post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Centering Guide Catheter
Number analyzed (Participants) | 20
Participants | 0

12. Other Pre Specified Outcome: Number of Device Deficiencies Including But Not Limited to Failures, Malfunctions, Use Errors, Product Nonconformities, and Labeling Errors
Description: All device deficiencies including but not limited to failures, malfunctions, use errors, product nonconformities, and labeling errors will be recorded in the case report form
Time Frame: 72 hours post-procedure
Measure: Count of Units; unit: Device
Units Other Than Participants: Device
Arm/Group | Self-Centering Guide Catheter
Number analyzed (Participants) | 20
Number analyzed (Device) | 23
Device | 1

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through 72 hours or discharge, whichever came first. There were no Adverse Events, Serious Adverse Events or Unanticipated Adverse Device Events, reported during the study period.
Arm/Group | Self-Centering Guide Catheter
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No